CLINICAL TRIAL: NCT05641311
Title: An Open-Label, Two-Single Dose, Two-Period, Parallel Group Study to Assess the Pharmacokinetics and Safety of ALXN1840 in Healthy Adult Japanese and Non-Japanese Subjects
Brief Title: Pharmacokinetic Study of Oral ALXN1840 in Japanese and Non-Japanese Adult Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WTX101-HV-106; 2018-004483-57 (EudraCT Number); C18055 (Other: RPL study code)
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Japanese Participants (Experimental): All Japanese participants will receive a single dose of ALXN1840 15 milligrams (mg) in Dosing Period 1 and will receive a single dose of ALXN1840 60 mg in Dosing Period 2.
  Interventions: Drug: ALXN1840
- Cohort 2: Non-Japanese Participants (Experimental): All non-Japanese participants will receive a single dose of ALXN1840 15 mg in Dosing Period 1 and will receive a single dose of ALXN1840 60 mg in Dosing Period 2.
  Interventions: Drug: ALXN1840

INTERVENTIONS:
Drug: ALXN1840 — Tablet for oral use.

SUMMARY:
The main purpose of the study is to confirm how long ALXN1840 stays in the body of Japanese and non-Japanese healthy participants (that is, pharmacokinetic [PK] profile).

ELIGIBILITY:
Key Inclusion Criteria: - Body weight ≤80 kilograms (kg) and body mass index (BMI) within the range 18-25 kg/m^2, inclusive, at screening. - Negative serum pregnancy test. - Female participants of childbearing potential and male participants with a female spouse or partner of childbearing potential must be willing to follow protocol-specified contraception guidance starting at least one menstrual cycle before first study drug administration and continuing for up to 3 months after the end of systemic exposure of the study drug (that is, 3 months after end of study visit).

Key Exclusion Criteria: - Current or recurrent/chronic disease (for example, cardiovascular, hematological, neurological, endocrine, immunological, rheumatological, renal, hepatic, or gastrointestinal (GI) or other conditions) that or could affect clinical assessments or clinical laboratory evaluations. - Current or relevant history of physical or psychiatric illness that are not stable or may require a change in treatment, use of prohibited therapies during the study or make the participant unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the study drug or study procedures. - Any other significant disease or disorder which, in the opinion of the Investigator, may put the participant at risk. - History of significant allergic reaction (for example, anaphylaxis or angioedema) to any product (for example, food, pharmaceutical). - Use of prescription medications (excluding oral contraceptives) within 14 days prior to dosing on Day 1, except with prior approval of Alexion. - Use of non-prescription/ over-the-counter medications including vitamins and dietary or herbal supplements, within 7 days prior to dosing on Day 1. - Donated or lost 400 milliliters (mL) blood or more within the last 16 weeks preceding the first day of dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Richmond Pharmacology Ltd., St George's University of London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For this study, Japanese participants were defined as those whose parents and grandparents were both Japanese and who had spent less than 5 years outside of Japan.
Pre-assignment Details: A total of 24 participants were screened, all of whom were enrolled and received ALXN1840 in the study at 1 study site. Of the 24 enrolled, 12 were Japanese, therefore, they were allocated to Cohort 1, and 12 were non-Japanese, therefore, they were allocated to Cohort 2. All participants were included in all analysis sets.
Groups:
- Cohort 1: Japanese Participants: All Japanese participants received a single dose of ALXN1840 15 milligrams (mg) in Dosing Period 1 and received a single dose of ALXN1840 60 mg in Dosing Period 2.
- Cohort 2: Non-Japanese Participants: All non-Japanese participants received a single dose of ALXN1840 15 mg in Dosing Period 1 and received a single dose of ALXN1840 60 mg in Dosing Period 2.
Period: Dosing Period 1
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Non-Japanese Participants
Started | 12 | 12
Received At Least 1 Dose Of Study Drug | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Dosing Period 2
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Non-Japanese Participants
Started | 11 | 12
Received At Least 1 Dose Of Study Drug | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all participants who received at least 1 dose of the study drug.
Groups:
- Cohort 1: Japanese Participants: All Japanese participants received a single dose of ALXN1840 15 mg in Dosing Period 1 and received a single dose of ALXN1840 60 mg in Dosing Period 2.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Non-Japanese Participants | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (5.91) | 29.5 (6.78) | 30.6 (6.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 1 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 11 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under The Plasma Concentration Versus Time Curve From Time 0 (Dosing) To The Last Quantifiable Concentration (AUCt) Of Plasma Total Molybdenum After Each Dose
Time Frame: Day 1 through Day 11 of Dosing Periods 1 and 2
Population: The PK population consisted of all participants who had sufficient plasma samples to enable the calculation of PK parameters of at least area under the curve (AUC) for at least one period.
Measure: Mean (Standard Deviation); unit: hours* nanograms/milliliters
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Non-Japanese Participants
Number analyzed (Participants) | 12 | 12
hours* nanograms/milliliters
  Dosing Period 1: ALXN1840 15 mg | 10158.9753 (1427.41833) | 9221.0132 (3413.75213)
  Dosing Period 2: ALXN1840 60 mg | 16178.7885 (6103.53245) | 20911.3717 (11491.5869)

ADVERSE EVENTS:
Time Frame: Baseline up to end of study visit (up to Day 29)
Description: The safety population consisted of all participants who received at least 1 dose of the study drug. All-Cause Mortality, Serious Adverse Event, and Other Adverse Event data were prespecified to be collected by their assigned cohort, regardless of their dose level.
Groups:
- Cohort 2: Non-Japanese Participants: All non-Japanese participants received a single dose of 15 mg ALXN1840 in Dosing Period 1 and a single dose of 60 mg ALXN1840 in Dosing Period 2.
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Non-Japanese Participants
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1: Japanese Participants (N=12) | Cohort 2: Non-Japanese Participants (N=12)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Medical device site reaction (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1/5 (1) | 0/5 (0) — The N for this adverse event has been adjusted to the number of females in the study as it is a sex-specific event.
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT05641311/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT05641311/SAP_001.pdf